CLINICAL TRIAL: NCT06992895
Title: Effect of Hologram Application on Pain, Anxiety and Fear Levels During Burn Dressing in Children: A Randomized Controlled Trial
Brief Title: Effect of Hologram Fan Application During Burn Dressing on Patient Comfort
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Muhammet MÜEZZİNOĞLU, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AU-HF-MM-01
Record Dates: First submitted 2025-04-25; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Burn Wounds; Burn
Keywords: Holography; Burns; Pain; Anxiety; Fear
MeSH Terms: conditions — Burns; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled trial.
Who Masked: Participant
Masking Description: Participants will be blinded by not being informed about the groups in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hologram fan group (Experimental): The technology of hologram fans will be employed in the 3D hologram fan group during the process of burn dressing. This technology utilizes LED lights to create three-dimensional visuals, thereby allowing children to draw their attention to different directions during dressing. Concurrently, scales designed to assess pain, anxiety, and fear will be completed during and immediately following the dressing process. The collection of data will be continued until the calculated number of participants is reached, as determined by the power analysis.
  Interventions: Device: The visual presentation utilizes a three-dimensional holographic fan device.
- Control group (No Intervention): The control group will be subjected to a state of distraction-free environment during the process of burn dressing. The group will undergo standard treatment procedures and will be treated exclusively with conventional methods. Concurrently, scales designed to assess pain, anxiety, and fear will be completed during and immediately following the dressing process. The collection of data will be continued until the calculated number of participants is reached, as determined by the power analysis.

INTERVENTIONS:
Device: The visual presentation utilizes a three-dimensional holographic fan device. — This study is among the first to examine the effect of holographic fan technology on pain, anxiety, and fear in children during burn dressing. In comparison with other distraction methods, holographic fans represent a novel technological intervention designed to mitigate pain and anxiety by engaging children's attention through the use of visual illusions. Furthermore, extant studies on the effectiveness of this technology during prolonged and distressing procedures, such as burn dressing, have been found to lack sufficient data.
  Arms: Hologram fan group

SUMMARY:
The process of dressing burn injuries has been shown to cause both physical and psychological difficulties. In children, this process is particularly associated with intense pain and anxiety. Consequently, in addition to pharmacological interventions, non-pharmacological methods such as distraction are employed. In recent years, the utilization of holograms as a method of alleviating pain has emerged as a novel approach. The employment of these visual illusions has been demonstrated to effectively distract children, thereby providing a means of reducing discomfort. The objective of this thesis is to evaluate the effects of hologram application on pain, anxiety, fear, and vital signs during burn dressing in children.

DETAILED DESCRIPTION:
Burns are defined as traumas caused by damage to the skin and subcutaneous tissues caused by heat, chemicals, electricity, or radiation. The severity of these injuries can range from superficial dermal damage to deep tissue loss. Burns inflict physical harm and can also cause significant psychological distress, including anxiety and fear, particularly in children. The administration of dressing procedures during the post-burn treatment process is a particularly challenging aspect for pediatric patients, often accompanied by significant anxiety and discomfort. Consequently, interventions that target both physical and psychological relaxation are necessary during the treatment process.

Among the technologies developed for the purpose of distraction in recent years, hologram fans are particularly noteworthy. The creation of three-dimensional visualizations by hologram fans utilizes LED lights strategically positioned on high-speed rotating propeller blades, resulting in the presentation of realistic images to the viewer, seemingly suspended in the air. This visual illusion has the potential to mitigate the discomfort and anxiety associated with medical procedures, particularly by capturing the attention of children. Research has demonstrated that the presence of hologram enthusiasts during pediatric medical procedures, such as blood draws, has been shown to reduce levels of fear and stress in children. However, the efficacy of these materials in applications requiring extended use and high levels of discomfort, such as burn dressings, remains to be adequately examined through scientific research.

This randomized controlled experimental study will examine the effect of a hologram fan application on pain, anxiety, and fear levels in pediatric burn patients receiving dressing changes. The study will be conducted with children between the ages of 3 and 12 who are receiving burn treatment in the hospital and require dressings. Those who meet the sampling criteria will be randomly assigned to the experimental or control group. The experimental group will receive a hologram fan display during dressing, while the control group will not receive any distracting method. Children in both groups will have their pain, anxiety, and fear levels measured before, during, and after dressing. Additionally, their basic vital signs, such as pulse and respiration, will be recorded during each dressing application.

ELIGIBILITY:
Inclusion Criteria:

* The subject has indicated their willingness to participate in the study. Physical and mental health.
* The age range of the subjects included in this study was from 3 to 12 years of age.
* The subject had never previously engaged in the practice of dressing a burn.
* The presence of only second degree burns
* Burn percentage is under 10%

Exclusion Criteria:

* The subject is unwilling or unable to provide informed consent or assent (if applicable).
* The subject has a history of significant physical or mental health disorders that may interfere with participation in the study.
* The subject is younger than 3 years old or older than 12 years old.
* The subject has previously engaged in the practice of burn dressing or similar procedures.
* The presence of burns other than second-degree burns (e.g., first-degree or third-degree burns).
* The percentage of burn area is greater than 10%.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The Wong-Baker Faces Pain Rating Scale: | up to 1 hours
  Measures the pain levels of children by describing their facial expressions. There are six different facial expressions, the lowest score is 0 and the highest score is 5.

SECONDARY OUTCOMES:
Children's Fear Scale (CFS): | up to 1 hours
  The level of fear is measured based on the change in facial muscle movements in children at the time of fear. The lowest score is 0 and the highest score is 4.

OTHER OUTCOMES:
State-Trait Anxiety Inventory for Children /STAI-CH): | up to 1 hours
  The State Anxiety Scale for Children is a self-report scale that evaluates children's momentary anxiety levels. The scale evaluates state anxiety based on emotions such as nervousness, tension, and uneasiness, and measures children's anxiety levels between 20 and 60 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Provincial Health Directorate Erzurum City Hospital, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No